CLINICAL TRIAL: NCT05509062
Title: Establishing Guidelines for Manual Lymphatic Drainage
Acronym: MLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0733
Record Dates: First submitted 2022-07-24; First posted 2022-08-19 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Lymphedema of Leg
MeSH Terms: interventions — Pressure

STUDY DESIGN:
Intervention Model Description: Treatment Group 1 Treatment Group 2 Treatment Group 3
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Light Tactile Pressure (Active Comparator): light tactile pressure with 5-10 mmHg without skin stretch
  Interventions: Procedure: Pressure
- Medium Tactile Pressure (Active Comparator): medium tactile pressure of 11-20 mmHg and medium skin stretch with therapist in a stationary position
  Interventions: Procedure: Pressure
- Firm Tactile Pressure (Active Comparator): firm tactile pressure (> 21 mmHg) and maximal skin stretch with therapist weight shift
  Interventions: Procedure: Pressure

INTERVENTIONS:
Procedure: Pressure — Subjects are randomized to one of three treatment groups

SUMMARY:
The purpose of this study is to establish optimal guidelines for Manual Lymphatic Drainage in participants with lower extremity lymphedema.

DETAILED DESCRIPTION:
To determine if there is a difference in L-Dex Score and Segmental Limb Volume in participants with lower extremity lymphedema as measured in liters by the SOZO machine between participants who receive Manual Lymphatic Drainage (MLD) techniques utilizing light tactile pressure with 5-10 mmHg without skin stretch versus medium tactile pressure of 11-20 mmHg and medium skin stretch with therapist in a stationary position, versus firm tactile pressure (> 21 mmHg) and maximal skin stretch with therapist weight shift.

ELIGIBILITY:
Inclusion Criteria:

* All adults between the age of 30 - 75 years
* Lower extremity lymphedema

Exclusion Criteria:

* Pregnant women
* Participants who are unable to stand independently for up to 2 mins
* Participants who cannot make their own decisions
* Participants undergoing cancer treatment
* Participants with an Infection (active cellulitis)
* Participants with a known Iodine Allergy
* Participants who weigh more than 375 lbs
* Participants with cardiac arrhythmias or implanted electronic equipment
* Participants who have undergone joint replacement in involved extremity
* Participants with cardiac insufficiency

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in The L-dex (Lymphedema Index). | 18 months
  The L-DEX score represents the difference in the amount of extracellular fluid in an at-risk limb compared to an unaffected limb.

SECONDARY OUTCOMES:
Change in Total body weight in liters | 18 Months
  All the water within a person's body, including both intracellular and extracellular fluid. Expressed as volume (liters or pints) and percentage of total weight (%).
Change in Extracellular Fluid in liters | 18 months
  All fluid that is not contained within the cells. Expressed as volume (liters or pints) and percentage of TBW (%).
Change in Intracellular Fluid in liters | 18 Months
  • Description: All fluid contained within the cells. Expressed as volume (liters or pints) and percentage of TBW (%).
Change in Skeletal Muscle Mass in lbs | 18 Months
  The amount of mass a person has that is made up of fat. Expressed in kgs or lbs and percentage of total weight (%)
Change in Fat Mass in lbs | 18 Months
  The amount of mass a person has that is made up of fat. Expressed in kgs or lbs and percentage of total weight (%)
Change in Free Fat Mass in lbs | 18 Months
  The amount of mass a person has that contains no fat (lean body mass). Includes muscle, connective tissue, organs, body water and bone. Expressed in kgs or lbs and percentage of total weight (%).
Change in Basal Metabolic Rate (BMR) in lbs | 18 Months
  Daily amount of energy a person's body burns when at complete rest. Expressed in calories.
Change in Basal Metabolic Rate in kg/m^2 | 18 months
  A relationship between weight and height that is associated with body fat and health risks. BMI = weight / height2.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Del Chiaro, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No